CLINICAL TRIAL: NCT00351832
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study to Compare the Effect of 12 Weeks Treatment With Vildagliptin (50mg qd, 50mg Bid, 100mg qd) to Placebo in Patients With Type 2 Diabetes
Brief Title: A Study To Compare the Effect of Vildagliptin Compared to Placebo in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A1303
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2007-05-09 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Vildagliptin; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study is not being conducted in the United States. Vildagliptin is an oral antidiabetic agent. This 12-week clinical study is to evaluate the effect of vildagliptin 50mg qd, 50mg bid or 100mg qd compared to placebo in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Patients who have been placed on dietary therapy/exercise therapy without achievement of glycemic control
* Outpatients

Exclusion Criteria:

* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes
* Significant cardiovascular disease
* Significant diabetic complications

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 236
Dates: Start 2006-06

PRIMARY OUTCOMES:
Change from baseline on HbA1c at 12 weeks

SECONDARY OUTCOMES:
Change from baseline on fasting plasma glucose at 12 weeks
Change from baseline on HOMA B at 12 weeks
Change from baseline on HOMA IR at 12 weeks
Change from baseline in body weight at 12 weeks
Change from baseline on fasting lipids at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan